CLINICAL TRIAL: NCT06647316
Title: The Effect of a Physioterapy Program on the Emotional Well-being of Patiens Admitted to an Acute Hospitalization Unit
Brief Title: Effects of an Early Physioterapy Program on the Emotional Well-being in Acute Hospitalized Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sierra Varona SL (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0014; 5607 (Registry Identifier: CEIm Hospital Universitario La Princesa)
Record Dates: First submitted 2024-10-11; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Acute Illness
Keywords: Well-being; Physiotherapy; Biopsychosocial Health Impact; Hospitalization
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: This project employs a quasi-experimental, analytical, longitudinal, prospective, single-group study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group: Physiotherapy for Emotional Well-Being (Experimental): The subjects will receive a minimum of four physiotherapy sessions in the various units where they are currently undergoing treatment. The treatment will be tailored to the specific pathology of each patient, in accordance with medical guidelines.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — The subjects will receive the first physiotherapy session : early mobilization, postural and joint ergonomics, sensory stimulation, temporal-spatial orientation and health education for the patient and the main caregiver are carried out.The plan will progress with postural control in a seated position, head and trunk control, re-education of transfers, balance, standing and walking, depending on the subject's abilities.The second physical therapy session incorporates taste and preference-based elements into the therapy itself. The third physiotherapy session is planned to take place in the physiotherapy unit. Following the individualized session, group interaction is encouraged, whether with other patients, the rehabilitation team and/or the patient's primary caregiver.In the fourth physiotherapy session, it is promoted therapeutic compliance.

SUMMARY:
Hospitalization due to acute illness often leads to a decline in physical function and quality of life, which significantly impacts the emotional well-being of patients, their families, and primary caregivers. Emotional well-being is a critical aspect of overall health, enabling individuals to cope with and adapt to health challenges. Addressing this dimension within the hospital setting is vital to improving patient outcomes, particularly from a biopsychosocial perspective that considers physical, psychological, and social factors.

This study aims to evaluate the effectiveness of physiotherapy interventions in enhancing the emotional well-being of hospitalized patients. While early physiotherapy is well-documented for its benefits in preventing complications and improving physical recovery, there is limited research demonstrating its impact on emotional well-being. Furthermore, data on the effects of prolonged hospitalization on the biopsychosocial health of patients is lacking.

Conducted at the Hospital Universitario de la Princesa (Madrid, Spain), a high-complexity hospital, this project will assess the role of physiotherapy not only in physical recovery but also in fostering emotional support. The intervention is designed to provide both therapeutic and emotional benefits, incorporating moments of relaxation and leisure into the treatment sessions. The study aligns with the growing global trend towards person-centered care and the humanization of healthcare.

This approach emphasizes a more holistic and personalized patient experience, where physiotherapy contributes to the overall health and well-being of the patient, addressing their physical and emotional needs.

DETAILED DESCRIPTION:
Background:

Hospitalization due to acute illness frequently results in a decline in physical function and quality of life, significantly affecting the emotional well-being of patients, their families, and primary caregivers. Emotional well-being is a crucial aspect of overall health, enabling individuals to cope with and adapt to health challenges. It is therefore essential that emotional well-being be addressed within the hospital setting if patient outcomes are to be improved, particularly from a biopsychosocial perspective that considers physical, psychological, and social factors.

The hypothesis is that the proposed intervention, which focuses on patients admitted to the Hospital Universitario de la Princesa de la Comunidad de Madrid, will effectively evaluate the role of hospital physiotherapy in improving emotional well-being.

Although the advantages of early physiotherapy in preventing complications and enhancing physical recovery are well-documented, there is a paucity of research demonstrating its impact on emotional well-being. Furthermore, there is a dearth of data concerning the effects of prolonged hospitalization on patients' biopsychosocial health.

The primary objective of this study is to assess the effectiveness of a physiotherapy intervention on the emotional well-being of patients admitted to the Hospital Universitario de La Princesa.

Secondary objectives includes:

* Examining the impact of sociodemographic factors on the efficacy of physical therapy.
* Evaluating the influence of physical therapy on the quality of life of patients admitted to the hospital.
* Analyzing the needs of the primary caregiver of admitted patients. It is hypothesized that physical therapy intervention in admitted patients at the Hospital Universitario de La Princesa improves their emotional well-being and quality of life.

Sample Recruitment Participants will be recruited through the rehabilitation physician, who also serves as the collaborating researcher and enrolls patients in the treatment program. Patients can be referred by the different medical services of the Hospital Universitario de la Princesa. Once a patient is enrolled in the study, a member of the research team will inform them of the study and provide them with the appropriate patient information sheet and informed consent form.

Study Design:

This project uses a quasi-experimental, analytic, longitudinal, prospective, single-group study design to examine the effects of a physical therapy intervention on the emotional well-being of inpatients. It employs a quasi-experimental design in which the investigator implements an intervention on a sample to examine the effects of physical therapy on emotional well-being and physical condition in real-world settings, with a focus on quality of life. This single-group pretest-posttest design involves assessing the same participants at two different points in time: before the physical therapy intervention begins (pretest) and after it ends (posttest).

Therapeutic intervention The subjects will receive the first physiotherapy session in the unit where they are currently being treated. The treatment will be adapted to the specific pathology of each patient, according to medical guidelines.

As a general intervention in immobilized patients, early mobilization, postural and joint ergonomics, sensory stimulation, temporal-spatial orientation and health education for the patient (according to the level of cooperation) and the main caregiver are carried out. The intervention is always adapted to the initial situation, pathology and needs.

According to the patient's progress, the treatment plan is modified after review by the rehabilitation physician in accordance with established guidelines. The plan will progress with postural control in a seated position, head and trunk control, re-education of transfers, balance, standing and walking, depending on the subject's abilities.

The second physical therapy session is also conducted at the patient's location within the unit, incorporating taste and preference-based elements into the therapy itself. This may include the ability to select the music to be played during the session. The individualized physiotherapy treatment is carried out according to the patient's pathology and in accordance with established medical guidelines. The goal is to promote the patient's physical autonomy in accordance with the current initial situation, using environmental indicators that facilitate the visualization of progress.

The third physiotherapy session is planned to take place in the rehabilitation gym, if the patient's clinical condition allows it. The same line of treatment will be continued and the humanizing approach developed on the ward will also be evident in the gym. Following the individualized session, group interaction is encouraged, whether with other patients, the rehabilitation team and/or the patient's primary caregiver.

If physical therapy is provided on the ward, it is also recommended that opportunities for group interaction with the professional team and/or primary caregiver be encouraged.

Group interaction will include the performance of activities in unison, including active mobility exercises for the upper and lower extremities, progressing to the administration of strengthening exercises for the primary muscle groups, and the implementation of therapeutic measures through the use of virtual reality glasses. The above-mentioned measures provide the patient with a calm, close and more humane therapeutic environment.

In the fourth physiotherapy session, a personalized element is introduced in the form of consumable materials provided by the service, with the aim of promoting therapeutic compliance and demonstrating the effort made by the patient.

The above procedures will be continued in the physiotherapy sessions throughout the patient's hospitalization.

Group interaction will include the performance of activities in unison, including active mobility exercises of the upper and lower extremities, followed by progressive strengthening exercises of the primary muscle groups. This will be done through the use of virtual reality goggles. The aforementioned measures are designed to provide the patient with a calmer, more intimate and more humane therapeutic environment.

Once the patient's clinical history is updated to indicate a probable discharge, the initial scales will be administered once more to both the patient and the caregiver. Furthermore, the patient will be provided with a questionnaire for the purpose of assessing satisfaction with the treatment received.

The physiotherapy intervention will comprise therapeutic exercises designed to facilitate physical recovery, while also integrating moments of relaxation and leisure into treatment sessions. This approach is aligned with the growing global trend toward person-centered care and the humanization of healthcare. It emphasizes a holistic and personalized patient experience, which is consistent with the principles of person-centered care and the humanization of healthcare.

Outcomes:

The primary outcome will be the assessment of emotional well-being, which will be measured using validated scales at two time points: before the intervention and after the intervention. Secondary outcomes will include assessments of physical function, quality of life, and patient satisfaction with the quality of care received.

Significance:

The objective of this study is to address the existing gap in the literature regarding the effectiveness of physiotherapy interventions on emotional well-being. By examining the impact of physiotherapy from a biopsychosocial perspective, this research aims to provide insights into the ways in which prolonged hospitalization affects patients' cognitive, social, and familial spheres. Moreover, it will highlight the necessity of integrating emotional support into physiotherapy practice

Clinical relevance:

The role of the physiotherapist is evolving to encompass not only the physical aspects of rehabilitation, but also the communication and emotional skills that facilitate optimal care. The findings of this study will contribute to the existing body of knowledge regarding the ways in which physiotherapy can enhance both physical and emotional recovery, thereby promoting a more comprehensive approach to patient care.

Etical and Legal Considerations:

This research project is conducted in accordance with all relevant ethical and legal regulations pertaining to research on human subjects.

This project will be conducted in accordance with the fundamental principles of Good Clinical Practice, as established in the Declaration of Helsinki and its subsequent modifications, the latest of which was the Fortaleza 2013 (World Medical Assembly), as set forth in the Council of Europe Convention on Human Rights and Biomedicine, and the UNESCO Universal Declaration on the Human Genome and Human Rights. Furthermore, the project will comply with the requirements set forth in the Spanish legislation pertaining to biomedical research, specifically the Law 14/2007 of July 3, 2007, on Biomedical Research and RD 1716/2011 on Biobanks, as well as the regulations concerning the protection of personal data.

ELIGIBILITY:
Inclusion Criteria:

-Volunteer Adults (18 years of age or older) that must provide written informed consent to participate in the study.

Hospitalization Requirements

* Participants must have been hospitalized in one of the hospital medical service departments for a minimum of 96 hours prior to enrollment.Eligibility for Physiotherapy:
* Participants must be deemed eligible for physiotherapy treatment during their hospital stay, as determined by the medical team.
* Cognitive Function: Participants must have a Mini-Mental State Examination (MMSE) score of 24 points or higher, indicating sufficient cognitive function.
* Participants must have received a minimum of 4 physiotherapy sessions during their hospital stay.
* A primary caregiver must be identified and available to participate in the study, although the caregiver does not need to be a family member.

Exclusion Criteria:

* Language Impairment: Patients with a language disorder that affects their ability to communicate effectively, thereby preventing them from providing informed consent or fully participating in the study.
* Language Barriers: Patients who encounter substantial linguistic barriers that cannot be overcome with the provision of interpretation or translation services, thus limiting their ability to comprehend or fully engage in the study.
* Patients Undergoing Specific Physiotherapeutic Treatments: Patients currently enrolled in physiotherapy programs standardized by the hospital's rehabilitation service for the following conditions: movement recovery, knee prosthesis, hip prosthesis, cardiac surgery, thoracic surgery, and bariatric surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Estimated)
Dates: Start 2024-10-14 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
WHO-5 Well-Being Index | The evaluation period will commence on the date of the initial documented progression and will conclude at least four days after the completion of the physical therapy sessions, or up to six days after the initial assessment.
  Emotional well-being will be assessed using the WHO-5 scale, a 5-item questionnaire that gathers ordinal qualitative data. Scores range from 0 to 25, where 25 represents the highest level of emotional well-being.

SECONDARY OUTCOMES:
EQ-5D-5L Scale | The evaluation period will commence on the date of the initial documented progression and will conclude at least four days after the completion of the physical therapy sessions, or up to six days after the initial assessment.
  Quality of life will be assessed using the EQ-5D scale, which covers five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain is scored using five response options, with higher scores indicating more unfavorable conditions. A visual analog scale (VAS) ranging from 0 to 100 will also be used to measure the patient's overall perception of health, where 100 represents optimal health.
Functional Ambulation Classification (FAC) Scale. Gait capacity | The evaluation period will commence on the date of the initial documented progression and will conclude at least four days after the completion of the physical therapy sessions, or up to six days after the initial assessment.
  Gait capacity will be evaluated using the FAC scale, which measures the degree of independence in walking. The scale consists of one item rated from 0 to 5, with 5 indicating the highest level of walking independence.
Critical Care Family Needs Inventory (CCFNI) | The evaluation period will commence on the date of the initial documented progression and will conclude at least four days after the completion of the physical therapy sessions, or up to six days after the initial assessment.
  The well-being of the family member or primary caregiver will be measured using the CCFNI, which consists of 14 items. The total score ranges from 14 to 56, with higher scores indicating worse outcomes.
Patient satisfaction: Study-Specific Questionnaire | The evaluation period will commence on the date of the initial documented progression and will conclude at least four days after the completion of the physical therapy sessions, or up to six days after the initial assessment.
  Patient satisfaction will be assessed using a 6-item questionnaire designed specifically for this study. Each item is rated on a scale of 1 to 5, with 5 indicating the highest level of satisfaction.

REFERENCES:
- [Background] Raurell-Torreda M, Arias-Rivera S, Marti JD, Frade-Mera MJ, Zaragoza-Garcia I, Gallart E, Velasco-Sanz TR, San Jose-Arribas A, Blazquez-Martinez E; Grupo MOviPre. Degree of implementation of preventive strategies for post-ICU syndrome: Multi-centre, observational study in Spain. Enferm Intensiva (Engl Ed). 2019 Apr-Jun;30(2):59-71. doi: 10.1016/j.enfi.2018.04.004. Epub 2018 Jun 28. English, Spanish. PMID 29960855
- [Background] Steenbruggen RA, Maas MJM, Hoogeboom TJ, Brand PLP, van der Wees PJ. A framework to improve quality of hospital-based physiotherapy: a design-based research study. BMC Health Serv Res. 2023 Jan 14;23(1):34. doi: 10.1186/s12913-023-09062-x. PMID 36641465
- [Background] Lobo A, Ezquerra J, Gomez Burgada F, Sala JM, Seva Diaz A. [Cognocitive mini-test (a simple practical test to detect intellectual changes in medical patients)]. Actas Luso Esp Neurol Psiquiatr Cienc Afines. 1979 May-Jun;7(3):189-202. No abstract available. Spanish. PMID 474231
- [Background] Cabases JM. [The EQ-5D as a measure of health outcomes]. Gac Sanit. 2015 Nov-Dec;29(6):401-3. doi: 10.1016/j.gaceta.2015.08.007. No abstract available. Spanish. PMID 26505321
- [Background] Holden MK, Gill KM, Magliozzi MR, Nathan J, Piehl-Baker L. Clinical gait assessment in the neurologically impaired. Reliability and meaningfulness. Phys Ther. 1984 Jan;64(1):35-40. doi: 10.1093/ptj/64.1.35. PMID 6691052
- [Background] Giordano A, Ferrari G, Radice D, Randi G, Bisanti L, Solari A; POSMOS study. Health-related quality of life and depressive symptoms in significant others of people with multiple sclerosis: a community study. Eur J Neurol. 2012 Jun;19(6):847-54. doi: 10.1111/j.1468-1331.2011.03638.x. Epub 2012 Jan 10. PMID 22233289

DOCUMENTS (1):
  • Informed Consent Form (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/16/NCT06647316/ICF_000.pdf